CLINICAL TRIAL: NCT05700968
Title: Investigation of the Validity and Reliability of the Turkish Version of Multidimensional Outcome Expectations For Exercise Scale (MOEES)
Brief Title: Turkish Version of Multidimensional Outcome Expectations For Exercise Scale (MOEES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yusuf Ziya Aarslan (Other)
Collaborators: İrem Hüzmeli (Unknown)
Responsible Party: Sponsor-Investigator, Yusuf Ziya Aarslan, Physiotherapist, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Other Study IDs: MKU-YZA-001
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Health Care Acceptor Health Knowledge, Attitudes, Practice Patient Participation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with cardiac disease
  Interventions: Other: validity and reability study

INTERVENTIONS:
Other: validity and reability study — Validity and reliability assessment of the Turkish version of the Multidimensional Outcome Expectations For Exercise Scale (MOEES).

SUMMARY:
The Multidimensional Outcome Expectations For Exercise Scale (MOEES) was developed to assess the multidimensional outcome expectations of exercise. The Turkish validity and reliability study of the scale, originally in English, has not been conducted before. The aim of this study is to develop the Turkish version of the Multidimensional Outcome Expectations For Exercise Scale (MOEES), and to report its reliability assessment.

DETAILED DESCRIPTION:
The Turkish version of The Multidimensional Outcome Expectations For Exercise Scale (MOEES) will be asked face to face with patients diagnosed with cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years.
* Be diagnosed with heart disease.
* Having at least one of the cardiac risk factors (hypertension, diabetes mellitus, hyperlipidemia/dyslipidemia, overweight or obesity (BMI>25), physical inactivity (less than 150 minutes of moderate-intensity exercise per week).
* To agree to participate in the study.
* Being able to write and speak in Turkish.

Exclusion Criteria:

* < 18 years.
* Lack of cooperation.
* No heart disease.
* Mental retardation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with cardiac disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2023-05-06 (Estimated); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
Reliability and Validity of MOEES by Correlation Analysis. | 6 months
  with MOEES will be researched

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia for Heart | 6 months
  The kinesiophobia levels of the patients will be evaluated.
International Physical Activity Questionnaire | 6 months
  The physical activity levels of the patients will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ziya Arslan, MSc., Principal Investigator — Mustafa Kemal University; İrem Hüzmeli, Dr., Study Director — Mustafa Kemal University

IPD SHARING:
Plan to Share IPD: Undecided